CLINICAL TRIAL: NCT00756418
Title: A Randomized Open-Label Comparative Study of Montelukast Versus Theophylline Added to Inhaled Corticosteroid in Pediatric Patients With Bronchial Asthma
Brief Title: Montelukast Post-marketing Comparative Study With Theophyline Added to Inhaled Corticosteroid (0476-396)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-396; MK0476-396; 2008_027
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Theophylline

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: montelukast
- 2 (Active Comparator)
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: montelukast — montelukast 5 mg QD 4-weeks.
  Other Names: MK0476
  Arms: 1
Drug: Theophylline — Theophylline 100 to 200 mg BID 4-weeks.
  Arms: 2

SUMMARY:
A clinical study explores the safety and efficacy of montelukast and to compare the safety and efficacy of montelukast with those of theophylline in pediatric bronchial asthma patients when they are used in conjunction with inhaled steroids.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Bronchial Asthma Patients Aged 6 To 14 Years (At The Beginning Of The Treatment Period)
* The Severity Must Be Mild, Moderate Or Severe, Persistent Bronchial Asthma
* The Patient Must Have Symptoms That Can Be Used As Efficacy Variables (Such As Repeated Coughing And Mild Or Moderate Asthma Attacks) During The Observation Period, And Must Be Using Inhaled Steroids

Exclusion Criteria:

* Patient Using Anti-Asthma Treatment Or Therapy Including corticosteroids Or Oral Anti-Allergic Drugs
* Patient With Complications That Will Impair The Judgment Of Efficacy Of This Drug
* Patient With Convulsive Disorders Such As Epilepsy Or Such A History
* Patient With Liver Disease, Renal Impairment, Heart Disease Or Such Other Complication

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2003-06-01 (Actual); Primary Completion 2004-08-28 (Actual); Study Completion 2004-08-28 (Actual)

PRIMARY OUTCOMES:
Improvement of AM PEF over first 2 Weeks | Over first 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kondo N, Katsunuma T, Odajima Y, Morikawa A. A randomized open-label comparative study of montelukast versus theophylline added to inhaled corticosteroid in asthmatic children. Allergol Int. 2006 Sep;55(3):287-93. doi: 10.2332/allergolint.55.287. PMID 17075269